CLINICAL TRIAL: NCT03497351
Title: Effects of Different Kinds of Antihypertensive Drugs on Dynamic Hemodynamic Changing of During Laparoscopic Gastrectomy and Laparotomy
Brief Title: Effects of Different Kinds of Hypotensive Drugs on Dynamic Hemodynamic Changing in Patients Under Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yi Liu, Attending doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: PLAGHAOC004
Record Dates: First submitted 2018-03-28; First posted 2018-04-13 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: General Surgery
MeSH Terms: interventions — Nicardipine; urapidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Experimental): the group treated with nicardipine
  Interventions: Drug: Nicardipine
- Group U (Experimental): the group treated with Urapidil
  Interventions: Drug: Urapidil

INTERVENTIONS:
Drug: Nicardipine — The patients in Group N were infused the 130/0.4 hydroxyethyl starch and sodium chloride injection ( 7 ml/kg, 0.4 ml/kg/min) after anesthesi induction and before skin incision. Then the HR, SAP, DAP, MAP, CO, CI, SV, SVI, PPV and SVV were recorded. When the circulation was stability, Nicardipine was given, and the the 130/0.4 hydroxyethyl starch and sodium chloride injection was infused again.
  Arms: Group N
Drug: Urapidil — The patients in Group N were infused the 130/0.4 hydroxyethyl starch and sodium chloride injection ( 7 ml/kg, 0.4 ml/kg/min) after anesthesi induction and before skin incision. Then the HR, SAP, DAP, MAP, CO, CI, SV, SVI, PPV and SVV were recorded. When the circulation was stability, Urapidil was given, and the the 130/0.4 hydroxyethyl starch and sodium chloride injection was infused again.
  Arms: Group U

SUMMARY:
SVV is clinically affected by a variety of factors, such as abdominal pressure, body position, tidal volume, type and temperature of liquid treatment, etc. There are few reports on the effects of drugs on SVV.

In clinical anesthesia, surgical stimulation and stress can affect patient hemodynamic stability, used in intraoperative vascular active drug is inevitable, they shrink or dilate blood vessels, speed up or slow down the heart rate, makes the ventricular preload and corresponding changes in the SV. Now, there is a study on SVV and PPV in patients with hypertension, but there are few reports on the effect of blood pressure drugs on the changes in patients' threshold.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ-Ⅲ
2. body mass index (BMI) 18-26kg/m2.
3. Hypertension and non-hypertensive patients
4. diabetic no complications
5. no lung, liver, kidney and blood system diseases
6. preoperative examination is basically normal.

Exclusion Criteria:

* Any type of arrhythmia, intraoperative need for other vasoactive drug intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
SVV | The period between the begining of anesthesia and the end of operation.
  stroke volume variation

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Haidian, China